CLINICAL TRIAL: NCT01758341
Title: Endoscopic Radiofrequency Ablation for Malignant Biliary Obstruction
Brief Title: Radiofrequency Ablation for Malignant Biliary Obstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Werner Dolak, MD, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK 1837/2012
Record Dates: First submitted 2012-12-11; First posted 2013-01-01 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Biliary Tract Neoplasms
Keywords: Malignant biliary obstruction; Endoscopic radiofrequency ablation; Therapeutic endoscopy
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Malignant biliary obstruction (Experimental): All patients who underwent endoscopic radiofrequency ablation with the HabibTM EndoHBP as a treatment for malignant biliary obstruction in Austria between November 2010 and December 2012.
  Interventions: Procedure: Endoscopic radiofrequency ablation; Procedure: Endoscopic retrograde cholangiopancreatography (ERCP); Device: HabibTM EndoHPB catheter

INTERVENTIONS:
Procedure: Endoscopic radiofrequency ablation — Endoscopic radiofrequency ablation with the HabibTM EndoHBP catheter uses bipolar electrical energy for tissue coagulation and can be applied without any special patient preparation in the context of an endoscopic retrograde cholangiopancreatography (ERCP) examination to treat malignant biliary strictures.
Procedure: Endoscopic retrograde cholangiopancreatography (ERCP) — ERCP is used to guide the RFA-catheter under radiological control to the location of the malignant stricture.
Device: HabibTM EndoHPB catheter — Used to apply radiofrequency energy to the malignant biliary stricture (see also intervention "endoscopic radiofrequency ablation")

SUMMARY:
Biliary obstruction is importantly influencing quality of life and survival of patients suffering from primary or secondary bile duct malignancies. The aim of this retrospective data analysis is to evaluate endoscopic radiofrequency ablation (RFA) with the HabibTM EndoHBP catheter for the treatment of malignant biliary obstruction. RFA procedures performed in Austria so far will be analyzed with regard to feasibility and safety of the technique. Therefore, the following parameters will be assessed: (among others) technical failures during the RFA procedure, complications during the RFA procedure, hospital stay, adverse events during hospital stay and until first clinical control after discharge (an expected average of 4 weeks after RFA procedure), 30-day and 90-day mortality. The results of this study should help to better understand important aspects of biliary RFA which may positively influence future applications of this method.

DETAILED DESCRIPTION:
Introduction

Biliary obstruction is the most relevant life limiting factor in patients suffering from primary or secondary bile duct malignancies. Underlying tumors, such as extrahepatic cholangiocarcinoma (CCa) of Klatskin type, pancreatic adenocarcinoma or metastases of colorectal cancer, are often diagnosed at an advanced stage when presenting with biliary obstruction. This mostly restricts treatment strategies to palliative management. Within this setting the prevention of biliary complications like jaundice, cholangitis or cholangiosepsis is one of the therapeutic key factors to extend survival and maintain quality of life [De Groen, Skipworth]. Endoscopic stenting of the biliary tract is an easy and safe approach to restore biliary drainage [Smith]. Self-expanding metal stents are preferred to plastic stents because of the lower risk of stent occlusion [Kaassis, Soderlund]. In addition to stenting endoscopic therapies that directly affect the local tumor mass, have been developed within the past years. First of all, photodynamic therapy using different photosensitizers has shown promising results for the reduction of tumor size and maintenance of biliary drainage [Ortner, Zoepf]. However, the patient management for this treatment involving peri-interventional photosensitivity remains cumbersome.

Recently, an endoscopically applicable radiofrequency catheter for the biliary tract, the so called HabibTM EndoHBP catheter, was introduced into the market. It uses bipolar electrical energy for tissue coagulation and can be applied without any special patient preparation in the context of an endoscopic retrograde cholangiopancreatography (ERCP) examination. RFA is well known from transcutaneous applications, where it already proved to be effective as a treatment option for hepatocellular carcinoma or intrahepatic CCa [Minami]. The new HabibTM EndoHBP catheter was already evaluated ex vivo [Itoi] and showed promising results concerning safety and prevention of stent occlusion in the context of one small retrospective clinical study [Steel].

Primary objective

Feasibility and safety of endoscopic radiofrequency ablation with the HabibTM EndoHBP catheter for the treatment of malignant biliary obstruction

Study Design

Retrospective analysis of prospectively gained clinical data

Primary endpoint

Technical failures during the RFA procedure

Secondary endpoints

1. Complications during the RFA procedure
2. Hospital stay
3. Adverse events during hospital stay and unil first clinical control after discharge (an expected average of 4 weeks after RFA procedure)
4. 30-day and 90-day mortality

Study Population

All patients who underwent endoscopic radiofrequency ablation with the HabibTM EndoHBP as a treatment for malignant biliary obstruction between November 2010 and December 2012 in Austria.

Methods

Endoscopic examination report databases will be screened for "radiofrequency ablation" in the context of an "endoscopic retrograde cholangiopancreatography" to identify the mentioned study population. Examination reports, discharge letters and patient curves of the study patients will be screened to yield the following parameters:

* Demographics

  * Sex
  * Age at first RFA-intervention
* Underlying disease that led to malignant biliary obstruction

  * Type of underlying disease
  * Time from diagnosis to first RFA-intervention
  * Previous treatment attempts (chemotherapy, radiation therapy, photodynamic therapy)
* Procedure related parameters

  * Prior biliary stents (type, amount)
  * Date of RFA procedure
  * Amount of RFA-applications during the procedure (energy, time)
  * Technical failure of the RFA catheter during the RFA procedure (defined as any technical problem that hinders the satisfactory application of RFA)
  * Complications during the RFA procedure (defined as any adverse change from the subject's baseline condition, i.e. any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease which is considered to be clinically relevant by the physician, whether or not considered related to the medical device)
  * Stenting after the procedure (type, amount)
* Post-interventional parameters

  * Days of hospitalization after the RFA procedure
  * Adverse events during hospital stay and until first clinical control after discharge (an expected average of 4 weeks after RFA procedure) defined as any adverse change from the subject's baseline condition, i.e. any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease which is considered to be clinically relevant by the physician, whether or not considered related to the medical device
  * Survial status (dead/alive) at the time of the data collection
  * (Cause of death)
  * (Time between first RFA procedure and death)

Data processing will be done after pseudonymization using continuous patient identification numbers. All parameters will be assessed descriptively. For scaled parameters (e.g. age) median and range will be calculated, for nominal parameters (e.g. type of underlying disease) the proportions of sub-items will be reported. Mortality will be assessed creating a Kaplan Meyer curve. 30-day and 90-day mortality will be extrapolated from this curve. All data processing will be done with SPSS 19.0.

Risk/Benefit assessment

Due to its retrospective design this study does not inherit any risk for the study patients.

Expected impact and Outlook

The results of this study may help to better understand the feasibility and safety profile of endoscopic radiofrequency ablation with the HabibTM EndoHBP catheter with potential effects on future applications.

ELIGIBILITY:
All patients who underwent endoscopic radiofrequency ablation with the HabibTM EndoHBP as a treatment for malignant biliary obstruction in Austria between November 2010 and December 2012.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of RFA-procedures with technical failures | During the respective RFA-examination (an expected average of 1 hour)
  The technical feasibility in this study will be specified as ratio of all technically successful RFA-applications to all examinations in which RFA-use was intended. A RFA-application will be classified as technically successful if it is possible to introduce the RFA-catheter into the biliary system, place it adequately accross the malignant stricture, apply RFA-energy and withdraw the RFA-catheter after RFA-application.

SECONDARY OUTCOMES:
Number of patients with interventional complications | During the respective RFA-procedure (an expected average of 1 hour)
  Clinically relevant complications occuring during the use of RFA, defined as any adverse change from the subject's baseline condition, which is considered to be clinically relevant by the physician, whether or not considered related to the medical device (e.g. bleeding, perforation).

OTHER OUTCOMES:
Hospital stay | Inpatient stay after RFA-procedure (an expected average of 5 days)
  Duration of hospitalization after the performance of RFA.
Number of patients with Adverse events as a Measure of Safety and Tolerability | During hospital stay and until first clinical control after discharge (an expected average of 4 weeks after RFA procedure)
  Adverse events occuring within 30 days after the RFA-procedure, defined as any adverse change from the subject's baseline condition, i.e. any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease which is considered to be clinically relevant by the physician, whether or not considered related to the medical device.
Mortality | 30 days and 90 days after RFA-procedure (calculating 30- and 90-day mortality rate), assessed retrospectively by screening clinical reports (including death reports) of the study patients on average 1 year after RFA-procedure
  Deaths occuring within 30 and 90 days after the RFA-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Werner Dolak, MD, Principal Investigator — Medical University of Vienna, Department of Internal Medicine III, Division of Gastroenterologie and Hepatologie
Locations (1):
- Medical University of Vienna, Department of Internal Medicine III, Division of Gastroenterology and Hepatology, Vienna, Austria

REFERENCES:
- [Background] de Groen PC, Gores GJ, LaRusso NF, Gunderson LL, Nagorney DM. Biliary tract cancers. N Engl J Med. 1999 Oct 28;341(18):1368-78. doi: 10.1056/NEJM199910283411807. No abstract available. PMID 10536130
- [Background] Skipworth JR, Olde Damink SW, Imber C, Bridgewater J, Pereira SP, Malago M. Review article: surgical, neo-adjuvant and adjuvant management strategies in biliary tract cancer. Aliment Pharmacol Ther. 2011 Nov;34(9):1063-78. doi: 10.1111/j.1365-2036.2011.04851.x. Epub 2011 Sep 20. PMID 21933219
- [Background] Smith AC, Dowsett JF, Russell RC, Hatfield AR, Cotton PB. Randomised trial of endoscopic stenting versus surgical bypass in malignant low bileduct obstruction. Lancet. 1994 Dec 17;344(8938):1655-60. doi: 10.1016/s0140-6736(94)90455-3. PMID 7996958
- [Background] Kaassis M, Boyer J, Dumas R, Ponchon T, Coumaros D, Delcenserie R, Canard JM, Fritsch J, Rey JF, Burtin P. Plastic or metal stents for malignant stricture of the common bile duct? Results of a randomized prospective study. Gastrointest Endosc. 2003 Feb;57(2):178-82. doi: 10.1067/mge.2003.66. PMID 12556780
- [Background] Soderlund C, Linder S. Covered metal versus plastic stents for malignant common bile duct stenosis: a prospective, randomized, controlled trial. Gastrointest Endosc. 2006 Jun;63(7):986-95. doi: 10.1016/j.gie.2005.11.052. PMID 16733114
- [Background] Ortner ME, Caca K, Berr F, Liebetruth J, Mansmann U, Huster D, Voderholzer W, Schachschal G, Mossner J, Lochs H. Successful photodynamic therapy for nonresectable cholangiocarcinoma: a randomized prospective study. Gastroenterology. 2003 Nov;125(5):1355-63. doi: 10.1016/j.gastro.2003.07.015. PMID 14598251
- [Background] Zoepf T, Jakobs R, Arnold JC, Apel D, Riemann JF. Palliation of nonresectable bile duct cancer: improved survival after photodynamic therapy. Am J Gastroenterol. 2005 Nov;100(11):2426-30. doi: 10.1111/j.1572-0241.2005.00318.x. PMID 16279895
- [Background] Minami Y, Kudo M. Radiofrequency ablation of hepatocellular carcinoma: Current status. World J Radiol. 2010 Nov 28;2(11):417-24. doi: 10.4329/wjr.v2.i11.417. PMID 21179308
- [Background] Itoi T, Isayama H, Sofuni A, Itokawa F, Tamura M, Watanabe Y, Moriyasu F, Kahaleh M, Habib N, Nagao T, Yokoyama T, Kasuya K, Kawakami H. Evaluation of effects of a novel endoscopically applied radiofrequency ablation biliary catheter using an ex-vivo pig liver. J Hepatobiliary Pancreat Sci. 2012 Sep;19(5):543-7. doi: 10.1007/s00534-011-0465-7. PMID 22038500
- [Background] Steel AW, Postgate AJ, Khorsandi S, Nicholls J, Jiao L, Vlavianos P, Habib N, Westaby D. Endoscopically applied radiofrequency ablation appears to be safe in the treatment of malignant biliary obstruction. Gastrointest Endosc. 2011 Jan;73(1):149-53. doi: 10.1016/j.gie.2010.09.031. PMID 21184881